CLINICAL TRIAL: NCT04598009
Title: A Phase II Study of Binimetinib in Combination With Imatinib in Patients With Advanced KIT-Mutant Melanoma
Brief Title: Binimetinib and Imatinib for Unresectable Stage III-IV KIT-Mutant Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20863; NCI-2020-07748 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
Keywords: KIT-Mutant; Unresectable Melanoma; Melanoma
MeSH Terms: conditions — Melanoma | interventions — binimetinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (binimetinib, imatinib) (Experimental): Patients receive binimetinib PO BID on days 1-28 and imatinib PO QD on days 1-28. Cycles repeat every 28 days
  Interventions: Drug: Binimetinib; Drug: Imatinib

INTERVENTIONS:
Drug: Binimetinib — Taken orally (PO) twice a day (BID)
  Other Names: Binimetinib Oral; Mektovi; ARRY-162; MEK162
Drug: Imatinib — Taken orally (PO) once a day (QD)
  Other Names: Imatinib Mesylate

SUMMARY:
This phase II trial studies how well binimetinib and imatinib work in treating patients with stage III-IV KIT-mutant melanoma that cannot be removed by surgery (unresectable). Binimetinib and imatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving binimetinib and imatinib may help treat patients with KIT-mutant melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the overall response rate (ORR) of binimetinib plus imatinib in participants with advanced KIT-mutant melanoma.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of binimetinib plus imatinib in participants with advanced KIT-mutant melanoma.

II. To estimate efficacy and survival parameters in participants with advanced KIT-mutant melanoma treated with binimetinib plus imatinib.

III. To estimate efficacy in participants with advanced KIT-mutant melanoma treated with binimetinib plus imatinib.

EXPLORATORY OBJECTIVES:

I. To investigate association between changes in drug phosphorylated end products (p-KIT, p-MEK, p-ERK) and clinical response.

II. To investigate association between clinical response and baseline Neurofibromatosis 1 (NF1) and SPRED1 status.

III. To investigate pathologic correlates of acquired resistance. IV. To investigate whether NF1 and SPRED1 loss contribute to acquired resistance.

V. To generate participant-derived xenograft models. VI. To determine the relationship between clinical outcomes and clinicopathologic features including KIT exon mutated, melanoma subtype, melanoma primary site, race/ethnicity, prior treatment history including immune checkpoint inhibitor (ICI)-experienced versus (vs) - naive.

OUTLINE:

Participants receive binimetinib orally (PO) twice daily (BID) on days 1-28 and imatinib PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at day 30 and 100, and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Have histologically or cytologically confirmed melanoma
* Have unresectable Stage III or Stage IV melanoma, as per American Joint Committee on Cancer 8th edition guidelines, not amenable to local therapy
* Have measurable disease by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) criteria
* Have documentation of KIT-mutant melanoma by Clinical Laboratory Improvement Act (CLIA)-certified testing platform
* Participants have progressed on prior standard-of-care therapy, or would be ineligible for or unable to tolerate standard-of-care therapy, in the opinion of the treating Investigator
* For participants who have received prior ICI, the following is permitted:

  * Prior adjuvant or neoadjuvant ICI, if last dose administered at least 4 weeks prior to study drug start
  * Prior ICI for the treatment of unresectable/metastatic disease, if last dose administered at least 4 weeks prior to study drug start
* Absolute neutrophil count >= 1,500/microliter (mcL)
* Platelets >= 100,000/mcL
* Total bilirubin below normal institutional limits, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) =< 3 x institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase (SGPT)) =< 3 x institutional upper limit of normal
* Creatinine =< 1.5 x within institutional upper limit of normal OR creatinine clearance glomerular filtration rate (GFR) >= 50 mL/min calculated using the Cockcroft-Gault formula
* Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy, with undetectable viral load within 3 months of study drug start, are eligible for this trial
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Individuals with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate central nervous system (CNS)-specific treatment is not required prior to study start
* Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Imatinib and/or binimetinib may have teratogenic effects. Women of child-bearing potential (WOCBP) must agree to:

  * Use highly effective contraception to avoid pregnancy from screening through 30 days after the last dose of study drugs;
  * Refrain from donating ova during the study through 30 days after the end of systemic exposure to study drugs;
  * Inform her treating physician immediately should she become pregnant or suspect she is pregnant while she is participating in this study
* Sexually active men enrolled on this protocol must agree to:

  * Use a condom for the duration of study participation and through 90 days after the end of systemic exposure to study drugs;
  * Refrain from donating sperm during the study through 90 days after the end of systemic exposure to study drugs;
  * If the male participant has a partner that is a WOCBP, that partner should also use highly effective contraception for the duration of the study and through 90 days after the end of the male participant's systemic exposure to study drug
  * Inform his treating physician immediately should his partner become pregnant while he is participating in this study

Highly effective (i.e., failure rate <1% per year when used consistently and correctly) methods of contraception include:

* Complete abstinence from heterosexual intercourse
* Combined (estrogen and progesterone) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intra-uterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized male partner (provided the vasectomized male has received medical assessment of surgical success, and that the male is a female participant's sole sexual partner)

  * Ability to understand a written informed consent document, and the willingness to sign it
  * The participant is deemed by the Investigator to have the initiative and means to be compliant with scheduled visits, treatment plan, and study procedures

Exclusion Criteria:

* Has received systemic anti-cancer therapies within 3 weeks of study drug start, radiation within 2 weeks, antibody therapy within 4 weeks
* Has not recovered from adverse events due to prior anti-cancer therapy to =< grade 1 or baseline. Note: Stable chronic conditions (grade =< 2) that are not expected to resolve (such as neuropathy, myalgia, alopecia, prior therapy-related endocrinopathies) are exceptions and may enroll
* Is currently receiving any other investigational agents or has received an investigational agent within 14 days or within 5 half-lives of investigational agent (whichever is shorter), prior to start of study drugs
* Inability to swallow and retain study drugs
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of study drugs (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, complete small bowel resection), or recent (=< 3 months) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs
* Hypersensitivity to binimetinib or any of its excipients
* Hypersensitivity to imatinib or any of its excipients
* Concurrent neuromuscular disorder that is associated with elevated creatinine-kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity of hypercoagulability syndromes); history of retinal degenerative disease
* Impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty of stenting) < 6 months prior to screening;
  * Congestive heart failure requiring treatment (New York Heart Association grade >= 2);
  * Left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO);
  * Uncontrolled hypertension defined as persistent systolic blood pressure >= 150 mmHg or diastolic blood pressure >= 100 mmHg despite current therapy;
  * History of presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
  * Triplicate average baseline corrected QT (QTc) interval >= 480 msec
* Use of a prohibited medication (including herbal medications, supplements, or foods) that cannot be safely discontinued prior to the start of study treatment
* Patients on warfarin who cannot be safely transitioned to an alternative systemic anticoagulant
* History of thromboembolic or cerebrovascular events =< 12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli. Note: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks prior to study drug start. Note: Patients with thromboembolic events related to indwelling catheters or other procedures may be enrolled
* Pregnant women are excluded from this study because binimetinib and imatinib are small molecule inhibitors with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with binimetinib and/or imatinib, breastfeeding should be discontinued prior to study drug start
* Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient an inappropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to week 16
  Defined as complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST v1.1). The ORR at stages 1 and 2 will be estimated using the method of Whitehead, and the p-values for testing the null hypothesis at each stage will use the method of Koyama & Chen and 90% confidence interval will be reported.

SECONDARY OUTCOMES:
Proportion of participants with treatment-related adverse events (AE) | Up to 2 years
  Proportion of participants with treatment-related AEs greater than grad2 as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 will be reported by toxicity.
Median duration of response | Up to 2 years
  Will estimate the probability-of-being-in-response function, assuming time to response is exponentially distributed.
Progression-free survival (PFS) | Up to 2 years
  Participants with an objective response will be followed for survival from initiation of study treatment until date of disease progression or death from any cause
Overall survival (OS) | Up to 2 years
  Participants will be followed from initiation of study treatment until date of disease progression or death from any cause and estimated using the Kaplan-Meier method to estimate the survival rate (95% CI)
Clinical benefit rate (CBR) | Up to 2 years
  Defined as CR, PR, or stable disease (SD) >= 16 weeks by RECIST. CBR will be defined as the proportion of participants with CR, PR, or SD for >= 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Katy Tsai, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No